CLINICAL TRIAL: NCT00015340
Title: Buprenorphine/Nx Treatment of Heroin Dependence-A Compassionate Use Study
Brief Title: Buprenorphine/Naloxone in the Treatment of Heroin Dependence - 14
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York MDRU (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-5-0013-14; Y01-5-0013-14
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-08

CONDITIONS: Opioid Dependence; Substance-Related Disorders
Keywords: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

ARMS (1):
- Buprenorphine/Naloxone (Experimental)
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is the safety and efficacy of Buprenorphine/Naloxone in the treatment of opioid dependence. A compassionate use study.

DETAILED DESCRIPTION:
The objective of this study is to provide follow-up compassionate use treatment and evaluate long term safety and efficacy of a buprenorphine/naloxone combination tablet for opiate dependence treatment for subjects who have completed Cooperative Study 1008 A and B.

ELIGIBILITY:
Inclusion Criteria:

- Completion of Cooperative Study 1008 A/B

Exclusion Criteria:

- Significant medical or psychiatric illness. Non-compliance with study procedures in the Cooperative Study 1008 A/B

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 582 (Actual)
Dates: Start 1999-08; Primary Completion 2001-08 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Craving
Retention
Opioid withdrawal
Subjective rating

CONTACTS AND LOCATIONS:
Overall Officials: Paul Casadonte, M.D., Study Chair — New York VAMC
Locations (5):
- United States (5):
  - University of California, Los Angeles, California
  - VA Medical Center, Tampa, Florida
  - VA Medical Center, Hines, Illinois
  - New York VAMC, New York, New York
  - VA PUget Sound Helath Care System, Seattle, Washington